CLINICAL TRIAL: NCT02536300
Title: Dose Optimization Study of Idelalisib in Follicular Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Gilead has made the decision to close the study due to enrollment challenges
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-313-1580; 2015-000366-66 (EudraCT Number)
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — idelalisib

STUDY DESIGN:
Intervention Model Description: As of protocol amendment 5, the Idelalisib 100 mg arm is closed to enrollment.
Masking Description: Double-blind: Prior to protocol amendment 5; Open-label: Participants enrolled as of protocol amendment 5
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Idelalisib 150 mg BID (Experimental): Participants will receive idelalisib 150 mg twice daily continuously.
  For participants enrolled prior to protocol amendment 5: Based on the independent review committee (IRC) response assessment, participants may be discontinued from the study or may receive blinded or open-label idelalisib 150 mg twice daily.
  Interventions: Drug: Idelalisib
- Idelalisib 100 mg BID (Experimental): Participants will receive idelalisib 100 mg twice daily continuously. Based on the IRC response assessment, participants may either be dose escalated to open-label 150 mg twice daily or maintain blind and continue on idelalisib 100 mg twice daily.
  As of protocol amendment 5, enrollment to this arm has been closed.
  Interventions: Drug: Idelalisib
- Idelalisib 150 mg BID INT (Experimental): Participants will receive idelalisib 150 mg twice daily in 28-day cycles with 21 days on-treatment and 7 days off-treatment.
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib tablet administered orally
  Other Names: Zydelig®; GS-1101; CAL-101

SUMMARY:
The primary objective of this study is to establish a safe and effective dosing regimen of idelalisib in participants with relapsed or refractory follicular lymphoma (FL) who have no other therapeutic options.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of B-cell follicular lymphoma (FL), and grade limited to 1, 2, or 3a based on criteria established by the World Health Organization (WHO) 2008 classification of tumors of hematopoietic and lymphoid tissues
* Relapsed or refractory FL and have received at least 2 lines of prior therapy for FL and have no other available therapeutic options. Note: Rituximab maintenance is not routinely considered a separate line of therapy when it is given as part of the prior rituximab-containing regimen given over a number of cycles followed by maintenance. Rituximab monotherapy may be considered a separate line of therapy when disease relapse occurs between the initiation of rituximab monotherapy and the preceding line of therapy. If there are any ambiguities about eligibility, the site should consult with the medical monitor.
* Ann-Arbor Stage 2 (non-contiguous), 3, or 4 disease per Lugano Classification Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥ 1 lesion that measures ≥ 1.5 cm in the longest dimension (LD) and ≥ 1.0 cm in the longest perpendicular dimension (LPD) as assessed by positron emission tomography-computed tomography (PET-CT), computed tomography (CT) or magnetic resonance imaging (MRI)
* Required baseline central laboratory data in protocol.
* For female individuals of childbearing potential and male individuals of reproductive potential, willingness to use a protocol- recommended method of contraception
* Lactating females must agree to discontinue nursing
* Willing and able to comply with scheduled visits, drug administration plan, imaging studies, laboratory tests, other study procedures, and study restrictions including mandatory prophylaxis for Pneumocystis jirovecii pneumonia (PJP)

Key Exclusion Criteria:

* History of lymphoid malignancy other than FL (eg, diffuse large B-cell lymphoma)
* Known history of, or clinically apparent, central nervous system (CNS) lymphoma or leptomeningeal lymphoma.
* Known presence of intermediate- or high-grade myelodysplastic syndrome.
* Known history of serious allergic reaction including anaphylaxis or Stevens- Johnson syndrome/ toxic epidermal necrolysis
* History of a non-lymphoid malignancy except for protocol allowed exceptions
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of enrollment
* Known history of drug-induced liver injury, chronic active hepatitis B virus (HBV), chronic active hepatitis C virus (HCV), alcoholic liver disease, non-alcoholic steatohepatitis, cirrhosis of the liver, portal hypertension, primary biliary cirrhosis, or ongoing extrahepatic obstruction caused by cholelithiasis
* History of or ongoing drug-induced pneumonitis
* History of or ongoing inflammatory bowel disease
* Known human immunodeficiency virus (HIV) infection
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy, including systemic corticosteroids (> 10 mg prednisone or equivalent/day) with the exception of the use of topical, enteric, or inhaled corticosteroids as therapy for comorbid conditions and systemic steroids for autoimmune anemia and/or thrombocytopenia
* Concurrent participation in another therapeutic clinical trial
* Prior treatment with phosphatidylinositol 3-kinase (PI3K) inhibitors
* Cytomegalovirus (CMV): Ongoing infection, treatment, or specifically CMV antiviral prophylaxis within 28 days prior to the screening visits CMV test

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (66):
- Calvary Norht Adelaide Hosptial, Woodville South, South Australia, Australia
- Royal Victoria Regional Health Centre, Barrie, Canada
- Czechia (3):
  - Fakultni nemocnice Brno, Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakulni newmcince v Motole, Onkologicka klinika 2. LF UK a FN Motol, Prague
- France (8):
  - Centre Hospitalier d'Avignon-Hopital Henri Duffaut, Avignon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Saint Antoine, Paris
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Universaitaire de Poit iers-Pole Regional de Cancerlogie, Poitiers
  - Centre Hospitalier de Tours-Hopital Bretoneau Centre Regional de Cancerologie Henry Kaplan, Tours
  - Clinique Louis Pasteur, Vandoeuvre-lés-Nancy
- Israel (2):
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
- Italy (16):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - ASST Spedali Civili, Brescia
  - Ospedale Policlinico San Martino IRCCS-Clinica Ematologica, Genoa
  - Azienda Policlinico San Martino, Genova
  - Azienda Ospedaliera Cardinale G Panico di Tricase-Unita Operativa Complessa di Ematologia e TMO, Lecce
  - Azienda Ospedaliera Vito Fazzi Unita Operativa di Ematologia, Lecce
  - Instituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Dipartimento di Oncologia Medica, Meldola
  - IRCCS Ospendale San Raffaele, Milan
  - SCDU Ematologia e Terapie Cellulari Azienda Ospedaliera Ordine Mauriziano di Torino, Orbassano
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Azienda Unita Sanitaria Locale di Ravenna, U.O di Ematologia, Ravenna
  - Ospedale degli Infermi-Oncoematologia, Rimini
  - Fondazione Policlinico Tor Vergata-UOC Patologie Linfoproliferative, Rome
  - Ospedale S. Eugenio, Rome
  - Dipartimento di Ematologia ed Oncoematolgia - S.C Ematolgia, Torino
  - A.S.U. Integrata Santa Maria della Misericordia, Udine
- Poland (9):
  - Szpitale Wojewodzkie w Gdyni Sp. z o.o., Gdynia
  - PRATIA Onkologia Katowice, Katowice
  - Malopolskie Centrum Medyczne, Krakow
  - Wojewodzki Szpital Specjalistyczny w Legniicy, Legnica
  - Gabinety Lekarskie Hema, Lublin
  - Szpital Wojewodzki w Opolu Sp. z o.o., Opole
  - Instytut Hematologii i Transfuzjologii, Klinika Hematologii, Warsaw
  - Centrum Onkologii Instytut im.Marii Sklodowskiej Curie, Warsaw
  - Klinika Hematologii Nowotworow Kriwi i Transplantacji Szpiku, Wroclaw
- Spitalul Judetean de Urgenta "Dr. Constantin Opris" Baia Mare, Baia Mare, Romania
- Spain (17):
  - Hospital del Mar, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro de Alcantara, Cáceres
  - Institut Catala d'Oncologia Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital General Universiario Gregorio Maranon, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Genereal Universitario Morales Meseguer, Murcia
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Mutua Terrassa, Terrassa
  - CEIm-Regional De La Comunidad De Madrid, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- United Kingdom (8):
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - London North West University Healthcare NHS Trust, Harrow
  - Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Barts Health Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - St George's Hospital NHS Trust, London
  - The Pennine Acute Hospital NHS Trust, Oldham
  - Torbay and South Devon NHS Foundation Trust, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-313-1580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Canada, Europe, Israel, and the United Kingdom.
Pre-assignment Details: 145 participants were screened.
Groups:
- Idelalisib 150 mg BID: Participants received idelalisib 150 mg tablets, orally, twice daily (BID), continuously for up to maximum 33.5 months.
- Idelalisib 100 mg BID: Participants received idelalisib 100 mg tablets, orally, BID, continuously for up to maximum 63.6 months.
- Idelalisib 150 mg BID INT: Participants received idelalisib 150 mg tablets, orally, BID for 21 days and 7 days off-treatment (intermittent [INT] dosing schedule) in each 28-day cycle for up to maximum of 24.6 months.
Period: Overall Study
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Started | 47 | 27 | 22
Completed | 0 | 0 | 0
Not Completed | 47 | 27 | 22
Not completed — Investigator's Discretion | 17 | 11 | 2
Not completed — Progressive Disease | 11 | 7 | 6
Not completed — Study Terminated by Sponsor | 6 | 4 | 7
Not completed — Death | 7 | 0 | 5
Not completed — Withdrew Consent | 4 | 2 | 0
Not completed — Initiation of Non-study Specific Anti-cancer Therapy in the Absence of Progression | 1 | 2 | 1
Not completed — Enrolled but Never Treated | 0 | 0 | 1
Not completed — Non-compliance With Study Drug | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Idelalisib 150 mg BID: Participants received idelalisib 150 mg tablets, orally, BID, continuously for up to maximum 33.5 months.
- Idelalisib 150 mg BID INT: Participants received idelalisib 150 mg tablets, orally, BID for 21 days and 7 days off-treatment (INT dosing schedule) in each 28-day cycle for up to maximum of 24.6 months.
- Total: Total of all reporting groups
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT | Total
Number analyzed (Participants) | 47 | 27 | 21 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 14 | 11 | 45
  >=65 years | 27 | 13 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (13.0) | 62 (13.6) | 63 (11.6) | 64 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 8 | 44
  Male | 24 | 14 | 13 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 42 | 26 | 17 | 85
  Unknown or Not Reported | 4 | 1 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 42 | 25 | 18 | 85
  Race: Unknown or Not Reported | 4 | 1 | 2 | 7
  Race: Asian | 1 | 0 | 0 | 1
  Race: Black or African American | 0 | 0 | 1 | 1
  Race: Other or More Than One Race | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 10 | 5 | 4 | 19
  Poland | 8 | 6 | 4 | 18
  Spain | 8 | 4 | 6 | 18
  United Kingdom | 6 | 5 | 4 | 15
  France | 5 | 2 | 2 | 9
  Czechia | 4 | 3 | 1 | 8
  Israel | 4 | 0 | 0 | 4
  Australia | 0 | 2 | 0 | 2
  Canada | 1 | 0 | 0 | 1
  Romania | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as percentage of participants who achieve a partial response (PR) or complete response (CR). PR criteria: No evidence of new disease, a ≥50% decrease from baseline in sum of products of diameters (SPD) of index lesions, no increase in non-index disease, no increase in liver/spleen size and no new liver/spleen enlargement. Persistence of bone marrow involvement in a participant who meets other criteria for CR based on the disappearance of all nodal and extra-nodal masses. CR criteria: No evidence of new disease, regression of all index nodal lesions to normal size (≤1.5 cm in longest dimension (LD) for large nodes and ≤1.0 cm in LD, ≤1.0 cm in longest perpendicular dimension (LPD) for small nodes), regression to normal of all nodal non-index disease, disappearance of all detectable extra-nodal index and non-index disease, normal spleen and liver size, no new liver/spleen enlargement, morphologically negative bone marrow.
Time Frame: Randomization up to end of treatment (maximum duration: 73.5 months)
Population: Intent-to-Treat (ITT) analysis set included all participants who were randomized regardless of whether they received any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 47 | 27 | 22
percentage of participants | 38.3 [24.5 to 53.6] | 44.4 [25.5 to 64.7] | 40.9 [20.7 to 63.6]

2. Primary Outcome: Number of Participants With Grade 4 or Higher Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as 1 or both of any AEs leading to premature discontinuation of study drug, or any AEs with an onset date on or after the study drug start date and no later than the last exposure date after permanent discontinuation of the study drug. TEAEs severity was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Fatal. Participants were counted at the highest AE grade experienced.
Time Frame: First dose date up to 30 days after last dose of study drug (maximum 64.6 months)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 47 | 27 | 21
Participants | 15 | 12 | 8

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR: interval from first documentation of CR/PR to earlier of first documentation of disease progression (PD) by independent review committee (IRC)/death from any cause. PR:No evidence of new disease,≥50% decrease from baseline in SPD of index lesions,no increase in non-index disease, no increase in liver/spleen size,no new liver/spleen enlargement; Persistence of bone marrow involvement in participant who meets other CR criteria. CR: No evidence of new disease,regression of all index nodal lesions to normal size (large nodes:≤1.5 cm in LD;small nodes:≤1.0 cm in LD,≤1.0 cm in LPD), regression to normal of all nodal non-index disease,disappearance of all detectable extra-nodal index,non-index disease,normal spleen and liver size, no new liver/spleen enlargement; PD: New node of >1.5 cm or >1.0 to ≤1.5 cm in LD, >1.0 cm in LPD, new/unequivocal reappearance of resolved extra-nodal lesion,new non-index disease,increase by 50% in SPD of index lesions,LD of individual node/extra-nodal mass.
Time Frame: From first documentation of CR or PR until PD or death from any cause (maximum duration: 73.5 months)
Population: Participants in the ITT analysis set who achieved CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 18 | 12 | 9
months | 27.1 [7.7 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of events. | 18.0 [2.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | 5.7 [0.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events.

4. Secondary Outcome: Overall Response Rate (ORR) by Week 24
Description: ORR by Week 24 is defined as the percentage of participants who achieve a PR or CR by Week 24.
  PR criteria: No evidence of new disease, a 50% decrease from baseline in SPD of index lesions, no increase in non-index disease, no increase in liver/spleen size and no new liver/spleen enlargement. CR criteria: No evidence of new disease, regression of all index nodal lesions to normal size (≤1.5 cm in LD for large nodes and ≤1.0 cm in LD, ≤1.0 cm in LPD for small nodes), regression to normal of all nodal non-index disease, disappearance of all detectable extra-nodal index and non-index disease, normal spleen and liver size, no new liver/spleen enlargement, morphologically negative bone marrow.
Time Frame: First dose date up to Week 24
Population: Participants in the ITT analysis set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 47 | 27 | 22
percentage of participants | 36.2 [22.7 to 51.5] | 33.3 [16.5 to 54.0] | 27.3 [10.7 to 50.2]

5. Secondary Outcome: Number of Participants With Any TEAE, Grade 3 or Higher TEAEs, Serious TEAEs, Idelalisib-related TEAEs, TEAEs Leading to Interruption or Discontinuation of Idelalisib
Description: TEAEs were defined as 1 or both of any AEs leading to premature discontinuation of study drug, or any AEs with an onset date on or after the study drug start date and no later than the last exposure date after permanent discontinuation of the study drug. TEAEs severity was graded according to the NCI CTCAE version 5.0. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Fatal. Participants are counted at the highest AE grade experienced.
Time Frame: First dose date up to 30 days after last dose of study drug (maximum 64.6 months)
Population: Participants in the safety analysis set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 47 | 27 | 21
Participants
  Any TEAE | 45 | 26 | 19
  Grade 3 or Higher TEAEs | 41 | 25 | 12
  Serious TEAEs | 31 | 19 | 11
  Idelalisib-related TEAEs | 38 | 25 | 11
  TEAEs Leading to Interruption of Idelalisib | 32 | 18 | 6
  TEAEs Leading to Discontinuation of Idelalisib | 28 | 13 | 4

6. Secondary Outcome: Number of Participants With Clinically Significant Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormality was defined as an increase of at least 1 toxicity grade from baseline at any time postbaseline up to and including the date of last study drug dose plus 30 days. Laboratory abnormalities included hematology and serum chemistry parameters. Clinically significant laboratory abnormalities were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for severity as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), or Grade 4 (life threatening). The number of participants with any post-baseline abnormal laboratory value in Grade 1-4 categories are reported.
Time Frame: First dose date up to 30 days after last dose of study drug (maximum 64.6 months)
Population: Participants in the safety analysis set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 47 | 27 | 20
Participants
  Hematology: Grade 1 | 7 | 5 | 2
  Hematology: Grade 2 | 12 | 7 | 5
  Hematology: Grade 3 | 15 | 11 | 5
  Hematology: Grade 4 | 6 | 3 | 2
  Serum Chemistry: Grade 1: number analyzed (Participants) | 47 | 27 | 19
  Serum Chemistry: Grade 1 | 9 | 5 | 8
  Serum Chemistry: Grade 2: number analyzed (Participants) | 47 | 27 | 19
  Serum Chemistry: Grade 2 | 17 | 8 | 4
  Serum Chemistry: Grade 3: number analyzed (Participants) | 47 | 27 | 19
  Serum Chemistry: Grade 3 | 10 | 11 | 6
  Serum Chemistry: Grade 4: number analyzed (Participants) | 47 | 27 | 19
  Serum Chemistry: Grade 4 | 7 | 3 | 1

7. Secondary Outcome: Time to Onset of Adverse Events of Interest (AEIs)
Description: Time to onset of AEIs is defined as the interval (in months) from the start of idelalisib treatment to the first documentation of start of AEI. AEIs included grade ≥ 3 diarrhea/colitis, rash, febrile neutropenia, infection, and any grade of: Pneumonitis, bowel perforation, progressive multifocal leukoencephalopathy (PML), Pneumocystis jirovecii pneumonia (PJP), cytomegalovirus (CMV) infection, and organizing pneumonia.
Time Frame: First dose date up to 30 days after last dose of study drug (maximum 64.6 months)
Population: AEIs data was not collected for analysis.
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the interval (in months) from randomization to the earlier of the first documentation of PD by IRC or death from any cause. PD criteria: New node of >1.5 cm or >1.0 cm to ≤1.5 cm in LD, >1.0 cm in LPD, new/unequivocal reappearance of resolved extra-nodal lesion, new non-index disease, increase by 50% in SPD of index lesions, LD of individual node/extra-nodal mass.
Time Frame: Randomization up to PD or death from any cause (maximum duration: 73.5 months)
Population: Participants in the ITT analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 47 | 27 | 22
months | 9.8 [5.5 to 28.7] | 19.4 [13.9 to 23.3] | 8.3 [2.9 to 8.7]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval (in months) from randomization to death from any cause.
Time Frame: Randomization up to death from any cause (maximum duration: 73.5 months)
Population: Participants in the ITT analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 47 | 27 | 22
months | 28.7 [14.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | NA [23.3 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of events. | NA [13.9 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of events.

10. Secondary Outcome: Trough Plasma Concentration of Idelalisib
Time Frame: Predose on Day 1, Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 32, and 48
Population: Pharmacokinetic (PK) analysis set included participants who received at least 1 dose of study drug and had at least 1 sample with detectable drug concentration. Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 44 | 27 | 21
nanograms per milliliter (ng/ml)
  Day 1: number analyzed (Participants) | 43 | 27 | 21
  Day 1 | NA (NA) — Mean and Standard Deviation (SD) were not available as the values were below the level of quantitation. | NA (NA) — Mean and SD were not available as the values were below the level of quantitation. | NA (NA) — Mean and SD were not available as the values were below the level of quantitation.
  Week 2: number analyzed (Participants) | 44 | 25 | 17
  Week 2 | 683.68 (514.166) | 382.94 (352.842) | 636.35 (461.042)
  Week 4: number analyzed (Participants) | 38 | 23 | 18
  Week 4 | 623.64 (466.557) | 447.78 (356.971) | 94.14 (231.647)
  Week 6: number analyzed (Participants) | 34 | 23 | 15
  Week 6 | 581.20 (470.988) | 361.90 (248.996) | 596.80 (401.619)
  Week 8: number analyzed (Participants) | 32 | 21 | 14
  Week 8 | 655.16 (498.873) | 430.33 (477.877) | 77.66 (274.313)
  Week 10: number analyzed (Participants) | 25 | 22 | 15
  Week 10 | 616.05 (370.862) | 356.12 (372.557) | 387.40 (314.249)
  Week 12: number analyzed (Participants) | 27 | 21 | 16
  Week 12 | 630.56 (664.066) | 389.21 (466.104) | 272.44 (626.451)
  Week 16: number analyzed (Participants) | 26 | 20 | 15
  Week 16 | 729.23 (832.158) | 730.29 (936.798) | 111.67 (296.666)
  Week 20: number analyzed (Participants) | 22 | 19 | 14
  Week 20 | 525.91 (411.330) | 745.58 (841.105) | 107.34 (269.434)
  Week 24: number analyzed (Participants) | 19 | 17 | 12
  Week 24 | 460.74 (321.766) | 728.76 (760.391) | NA (NA) — Mean and SD were not available as the values were below the level of quantitation.
  Week 32: number analyzed (Participants) | 16 | 11 | 11
  Week 32 | 446.13 (450.821) | 388.58 (351.293) | 352.73 (875.923)
  Week 48: number analyzed (Participants) | 8 | 8 | 5
  Week 48 | 706.13 (580.022) | 552.13 (571.081) | 165.00 (368.951)

11. Secondary Outcome: Peak Plasma Concentration of Idelalisib
Time Frame: 1.5 hours postdose on Day 1, Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 32, and 48
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
Number analyzed (Participants) | 43 | 27 | 20
ng/ml
  Day 1 | 2626.12 (1330.290) | 1575.81 (803.317) | 2221.35 (1621.291)
  Week 2: number analyzed (Participants) | 42 | 24 | 18
  Week 2 | 2306.12 (810.433) | 1520.29 (675.089) | 2186.89 (1265.850)
  Week 4: number analyzed (Participants) | 39 | 23 | 17
  Week 4 | 2353.95 (930.754) | 1528.48 (759.936) | 2608.12 (1009.937)
  Week 6: number analyzed (Participants) | 30 | 21 | 15
  Week 6 | 2433.33 (1092.969) | 1682.52 (939.455) | 2341.33 (948.133)
  Week 8: number analyzed (Participants) | 29 | 20 | 14
  Week 8 | 2207.59 (980.606) | 1649.25 (940.683) | 2786.43 (1591.408)
  Week 10: number analyzed (Participants) | 24 | 19 | 15
  Week 10 | 2435.00 (1027.469) | 1601.11 (804.605) | 2380.00 (1118.679)
  Week 12: number analyzed (Participants) | 24 | 19 | 15
  Week 12 | 2328.13 (1141.764) | 1658.89 (837.159) | 2316.20 (1391.815)
  Week 16: number analyzed (Participants) | 23 | 20 | 12
  Week 16 | 2634.39 (1323.611) | 1756.37 (826.784) | 2372.50 (1335.420)
  Week 20: number analyzed (Participants) | 19 | 17 | 13
  Week 20 | 2354.26 (1440.587) | 1925.29 (776.516) | 2177.69 (1417.505)
  Week 24: number analyzed (Participants) | 15 | 17 | 10
  Week 24 | 2058.47 (905.071) | 1914.65 (1151.998) | 1906.30 (1099.458)
  Week 32: number analyzed (Participants) | 14 | 10 | 10
  Week 32 | 2009.71 (1231.296) | 2028.00 (593.236) | 1825.00 (947.892)
  Week 48: number analyzed (Participants) | 8 | 9 | 5
  Week 48 | 2655.13 (1348.957) | 1448.33 (650.798) | 1312.00 (850.894)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to last follow up visit (maximum 73.5 months); Adverse Events: First dose date up to 30 days after last dose of study drug (maximum 64.6 months)
Description: All-Cause Mortality: All enrolled analysis set included all participants who received a study participant identification number after screening and was used for participant enrollment summary and data listings, unless otherwise specified.
  Adverse Events: Safety analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | Idelalisib 150 mg BID | Idelalisib 100 mg BID | Idelalisib 150 mg BID INT
All-Cause Mortality (participants affected / at risk) | 20/47 | 12/27 | 6/22
Serious Adverse Events (participants affected / at risk) | 31/47 | 19/27 | 11/21
Other Adverse Events (participants affected / at risk) | 44/47 | 24/27 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib 150 mg BID (N=47) | Idelalisib 100 mg BID (N=27) | Idelalisib 150 mg BID INT (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0
Visual field defect (Eye disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 0
Facial pain (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Coronavirus pneumonia (Infections and infestations) | 1 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 1 | 2
Covid-19 pneumonia (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0
Klebsiella test positive (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 4 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib 150 mg BID (N=47) | Idelalisib 100 mg BID (N=27) | Idelalisib 150 mg BID INT (N=21)
Anaemia (Blood and lymphatic system disorders) | 10 | 3 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 10 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 2
Colitis (Gastrointestinal disorders) | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 19 | 12 | 6
Nausea (Gastrointestinal disorders) | 5 | 6 | 4
Vomiting (Gastrointestinal disorders) | 4 | 5 | 1
Asthenia (General disorders) | 4 | 4 | 3
Fatigue (General disorders) | 5 | 2 | 2
Oedema peripheral (General disorders) | 5 | 2 | 3
Pyrexia (General disorders) | 11 | 6 | 3
Bronchitis (Infections and infestations) | 2 | 1 | 2
Covid-19 (Infections and infestations) | 1 | 1 | 2
Influenza (Infections and infestations) | 3 | 0 | 0
Oral candidiasis (Infections and infestations) | 4 | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 0
Urinary tract infection (Infections and infestations) | 3 | 4 | 2
Alanine aminotransferase increased (Investigations) | 9 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 6 | 0
Transaminases increased (Investigations) | 1 | 0 | 2
Weight decreased (Investigations) | 4 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 3 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 4 | 6
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 5 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT02536300/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02536300/SAP_001.pdf